CLINICAL TRIAL: NCT00425672
Title: Phase I-II Study of Denileukin Diftitox (ONTAK®) in Patients With Advanced Refractory Breast Cancer
Brief Title: ONTAK® in Treating Patients With Advanced Breast Cancer That Did Not Respond to Previous Treatment
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Mary (Nora) Disis, Principal Investigator, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6308 (FH/UWCC ID); NCI-2010-00800 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 127 (Other: Tumor Vaccine Group); NCT00364208 (obsolete NCT alias)
Record Dates: First submitted 2007-01-19; First posted 2007-01-23 (Estimated); Results first posted 2017-08-04 (Actual); Last update posted 2018-12-05 (Actual); Status verified 2018-11

CONDITIONS: Male Breast Cancer; Recurrent Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer; Stage IV Breast Cancer
MeSH Terms: conditions — Breast Neoplasms, Male; Breast Neoplasms | interventions — denileukin diftitox; Flow Cytometry; Immunohistochemistry; Enzyme-Linked Immunosorbent Assay

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm I (Experimental): Patients receive ONTAK IV over 1 hour on days 1-5. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: ONTAK; Other: flow cytometry; Other: immunohistochemistry staining method; Other: enzyme-linked immunosorbent assay; Other: laboratory biomarker analysis; Genetic: protein expression analysis

INTERVENTIONS:
Biological: ONTAK — Given IV
  Other Names: DAB389 interleukin-2; DAB389 interleukin-2 immunotoxin; DAB389-IL2; DAB389IL-2; denileukin diftitox; DAB389IL2; DABIL2
Other: flow cytometry — Correlative studies
Other: immunohistochemistry staining method — Correlative studies
  Other Names: immunohistochemistry
Other: enzyme-linked immunosorbent assay — Correlative studies
  Other Names: ELISA
Other: laboratory biomarker analysis — Correlative studies
Genetic: protein expression analysis — Correlative studies

SUMMARY:
RATIONALE: ONTAK may be able to help reduce the type of cells that prevent other types of immune cells from attacking the breast cancer cells.

PURPOSE: This phase I/II trial is studying the safety of ONTAK and its possible side effects to see how well it works in treating patients with advanced breast cancer that did not respond to previous treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety of ONTAK infusion in patients with advanced refractory breast cancer.

II. To evaluate the effect of ONTAK administration on peripheral blood T-regulatory cells.

SECONDARY OBJECTIVES:

I. To evaluate the incidence of IL-2R expression in tumor samples and investigate the correlation of tumor IL-2R expression and tumor response to ONTAK therapy.

II. To evaluate levels of circulating sIL-2R before and after ONTAK therapy. III. To evaluate the effect of ONTAK on endogenous tumor specific immunity. IV. To evaluate the potential anti-tumor effects of ONTAK in patients with advanced refractory breast cancer.

OUTLINE:

Patients receive ONTAK IV over 1 hour on days 1-5. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced stage refractory breast cancer
* Progressive or relapsed disease following standard therapy
* Patients must have measurable disease that can include, but is not limited to bone; specifically, patients must have measurable extraskeletal disease that can be accurately measured in at least one dimension as >= 20 mm with conventional CT techniques or >= 10 mm with spiral CT scan; measurable (bi-dimensional) chest wall disease will also be allowed
* Patients must be at least 14 days out from last cytotoxic chemotherapy; patients on bisphosphonates are eligible
* White blood cell count (WBC) > 3.0 THOU/ul
* ANC > 1.0 THOU/ul
* Platelets >= 100 THOU/ul
* Serum creatinine =< 2.0 mg/dL or creatinine clearance (calculated) >= 60 ml/min
* ALT/AST =< 2.0 x upper limit of normal
* Total bilirubin =< 1.5 x upper limit of normal
* Albumin >= 3.0 g/dL
* Subjects must have a Performance Status Score (ECOG Scale) =< 2
* Subjects must have recovered from major infections and/or surgical procedures and, in the opinion of the investigator, not have a significant active concurrent medical illness precluding protocol treatment
* Men and women of reproductive ability must agree to contraceptive use during the study and for 1month after ONTAK treatment is discontinued

Exclusion Criteria:

* Prior treatment with ONTAK (DAB389 IL-2) or DAB486 IL-2
* Known history of hypersensitivity to diphtheria toxin or IL-2
* Active autoimmune disease
* Known history of pulmonary disease except controlled asthma
* History of or pre-existing, cardiovascular disease as defined by New York Heart Association (NYHA) Class III-IV categorization
* Pregnant or breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2005-09 (Actual); Primary Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lupe Salazar, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- ONTAK: Patients receive ONTAK IV over 1 hour on days 1-5. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  ONTAK: Given IV
  flow cytometry: Correlative studies
  immunohistochemistry staining method: Correlative studies
  enzyme-linked immunosorbent assay: Correlative studies
  laboratory biomarker analysis: Correlative studies
  protein expression analysis: Correlative studies
Period: Overall Study
Arm/Group | ONTAK
Started | 15
Completed | 14
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Arm I
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Safety Evaluated by Collecting Study Related Toxicity as Assessed by CTCAE v3.0
Description: Subjects are monitored for the development of end organ damage by assessing adverse events with serum chemistries, liver function studies, serum albumin, complete blood counts, symptom assessment, and physical exams performed at every cycle until 3 weeks after the final dose of ONTAK. All adverse events for all systems are graded on a scale of 1-5 using CTCAE v3.0.
Time Frame: 7 Days after last dose of ONTAK
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I
Number analyzed (Participants) | 15
Participants | 15

2. Primary Outcome: Efficacy of ONTAK in Depleting T-regulatory Cells as a Decrease in Peripheral Blood Tregs Using Flow Cytometry
Description: The efficacy of ONTAK in depleting Tregs will be defined as a decrease in peripheral blood Tregs by 25% of each individual subject's baseline. All subjects will undergo blood draws at baseline and post ONTAK infusions at designated time points. Tregs from the peripheral blood will be quantitated using flow cytometry.
Time Frame: 21 days after cycle 6
Population: 14 patients equals patients that had repeat blood draws taken but did not complete the treatment except for 4 patients who completed the study
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I
Number analyzed (Participants) | 14
Participants | 4

3. Secondary Outcome: Incidence of Interleukin-2 (IL-2) and IL-2 Receptor (IL-2R) Expression in Tumor Samples by Immunohistochemical (IHC) Analysis
Description: The incidence of IL-2 expression and its receptor complex, IL-2R in tumor samples will be evaluated by IHC analysis. Tumor sections will be interpreted as either positive or negative.
Time Frame: 21 days after cycle 6
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I
Number analyzed (Participants) | 14
Participants
  YES | 8
  NO | 6

4. Secondary Outcome: Presence of Circulating sIL-2R in the Peripheral Blood
Description: Evaluate levels of circulating sIL-2R (pg/ml) in the peripheral blood assessed before and after ONTAK therapy. Changes from baseline will be tabulated.
Time Frame: 21 days after cycle 6
Population: 4/14 patients had peripheral blood available before and after ONTAK treatment.
Measure: Median (Full Range); unit: pg/ml
Arm/Group | Arm I
Number analyzed (Participants) | 14
pg/ml
  Pre ONTAK Treatment: number analyzed (Participants) | 4
  Pre ONTAK Treatment | 4.8 [1.3 to 673.0]
  6 Weeks Post ONTAK Treatment | 8.1 [3.0 to 360.5]
  12-16 Weeks Post ONTAK Treatment | 34.8 [3.4 to 58.1]
  18-23 Weeks Post ONTAK Treatment | 17.7 [2.7 to 282.5]

5. Secondary Outcome: Presence of Endogenous Tumor-specific Immunity
Description: Evaluate the effect of ONTAK on endogenous tumor specific immunity
Time Frame: 21 days after cycle 6
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I
Number analyzed (Participants) | 14
Participants | 10

6. Secondary Outcome: Anti-tumor Effects of ONTAK Determined by Tumor Response and Progression
Description: Anti-tumor effects of ONTAK will be determined by evaluating tumor response and progression per RECIST. An objective response to ONTAK will be defined as achieving a CR or PR. Analysis of the data will include determination of complete (CR) and partial response (PR) rates, as well as stable (SD) and progressive disease (PD).
Time Frame: 21 days after cycle 6
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I
Number analyzed (Participants) | 15
Participants
  Complete Response (CR) | 0
  Partial Response (PR) | 0
  Progressive Disease (PD) | 10
  Stable Disease (SD) | 4

ADVERSE EVENTS:
Arm/Group | Arm I
Serious Adverse Events (participants affected / at risk) | 1/15
Other Adverse Events (participants affected / at risk) | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (N=15)
Severe Nausea and Vomiting (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (N=15)
Allergic Reaction/Hypersensitivity (Investigations) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Other - Ringing in Ear (Ear and labyrinth disorders) | 1 (1)
Hemoglobin Abnormal (Blood and lymphatic system disorders) | 8 (18)
Lymphopenia (Blood and lymphatic system disorders) | 4 (8)
Platelets Abnormal (Blood and lymphatic system disorders) | 3 (6)
Leukocytes Abnormal (Blood and lymphatic system disorders) | 2 (7)
ANC/AGC Abnormal (Blood and lymphatic system disorders) | 2 (3)
Blood and Lymphatic System Disorders - Other (Blood and lymphatic system disorders) | 1 (3) — RBC Low
Blood and Lymphatic System Disorders - Other (Blood and lymphatic system disorders) | 1 (1) — MCV and MCH High
Blood and Lymphatic System Disorders - Other (Blood and lymphatic system disorders) | 1 (2) — HCT Low
Cardiac Arrhythmia (Cardiac disorders) | 1 (2)
Hypotension (Vascular disorders) | 2 (4)
Hypertension (Cardiac disorders) | 1 (2)
Fatigue (General disorders) | 12 (36)
Rigors/Chills (General disorders) | 11 (12)
Insomnia (Psychiatric disorders) | 10 (14)
Fever (General disorders) | 4 (5)
Weight Gain (Gastrointestinal disorders) | 1 (2)
Weight Loss (Gastrointestinal disorders) | 1 (1)
Rash/Desquamation (Skin and subcutaneous tissue disorders) | 2 (2)
Rash: Acne/Acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Flushing (Vascular disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 12 (26)
Nausea (Gastrointestinal disorders) | 9 (22)
Anorexia (Gastrointestinal disorders) | 9 (14)
Vomiting (Gastrointestinal disorders) | 7 (10)
Diarrhea (Gastrointestinal disorders) | 4 (5)
Gastritis (Gastrointestinal disorders) | 2 (2)
Taste Alteration (dysgeusia) (Nervous system disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (2)
Infection - Toe (Infections and infestations) | 1 (1)
Edema: Limb (Vascular disorders) | 4 (6)
AST Abnormal (Investigations) | 14 (34)
ALT Abnormal (Investigations) | 14 (33)
Hypocalcemia (Metabolism and nutrition disorders) | 12 (28)
Hypoalbuminemia (Metabolism and nutrition disorders) | 11 (27)
Hypokalemia (Metabolism and nutrition disorders) | 10 (31)
Hyperglycemia (Metabolism and nutrition disorders) | 8 (21)
Creatinine Abnormal (Metabolism and nutrition disorders) | 8 (19)
Alkaline Phosphatase Abnormal (Investigations) | 6 (11)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (4)
Hypoproteinemia (Investigations) | 2 (7)
Hyponatremia (Metabolism and nutrition disorders) | 1 (2)
Alkalosis (metabolic or respiratory) (Metabolism and nutrition disorders) | 1 (1)
Hyperbilirubinemia (Metabolism and nutrition disorders) | 1 (1)
Chloride High (Metabolism and nutrition disorders) | 1 (5)
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1 (2)
Leg Cramps (Metabolism and nutrition disorders) | 1 (1)
Dizziness (Nervous system disorders) | 4 (5)
Neuropathy: Sensory (Nervous system disorders) | 4 (4)
Mood Alteration (Psychiatric disorders) | 3 (3)
Confusion (Psychiatric disorders) | 2 (2)
Ataxia (incoordination) (Nervous system disorders) | 1 (1)
Neuropathy: Motor (Nervous system disorders) | 1 (4)
Loss of Acuity Related to Illness (Eye disorders) | 1 (1)
Vitreous Detachment (Eye disorders) | 1 (1)
Vision Blurred - Vision (Eye disorders) | 1 (1)
Watery Eye (Eye disorders) | 1 (1)
Headache (Nervous system disorders) | 10 (18)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (8)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (6)
Pain - Chest Wall (Musculoskeletal and connective tissue disorders) | 4 (4)
Pain - Back (Musculoskeletal and connective tissue disorders) | 3 (7)
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 3 (3)
Pain - Bone (Musculoskeletal and connective tissue disorders) | 2 (3)
Abdomen NOS (Gastrointestinal disorders) | 2 (3)
Extremity (Musculoskeletal and connective tissue disorders) | 1 (2)
Pain - Arm (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain - Musculoskeletal - Extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain - Rib (Musculoskeletal and connective tissue disorders) | 1 (1)
Throat/Pharynx/Larynx (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain - Tightness in Shoulders Secondary to Benadryl IV (General disorders) | 1 (1)
Dyspnea (Shortness of Breath) (Respiratory, thoracic and mediastinal disorders) | 9 (11)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (12)
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Pleural Effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary Fibrosis (radiologic changes) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Flu-Like Syndrome (General disorders) | 5 (10)
Acute Vascular Leak Syndrome (Vascular disorders) | 10 (19)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes